CLINICAL TRIAL: NCT06833723
Title: Construction and Validation of a Multi-omics Prediction Model to Assess Immunotherapy Efficacy in Patients With Triple-Negative Breast Cancer Subtypes Based on Genomic, Transcriptomic, Proteomic, and Immune Profiling Data
Brief Title: Development of a Multi-omics Prediction Model for Immunotherapy Response in Triple-Negative Breast Cancer Subtypes
Status: Active, not recruiting | Type: Observational
Sponsor: Hangzhou Institute of Medicine (HIM), Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, Qin Wu, Research Professor, Hangzhou Institute of Medicine (HIM), Chinese Academy of Sciences
Other Study IDs: HIM-1
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — * Fresh tumor biopsy samples preserved in RNAlater solution for proteomics and transcriptomics sequencing.
  * Fresh frozen samples stored at -80°C for imaging mass cytometry and spatial transcriptomics analysis.
  * Blood samples collected for metabolomics sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort (2015-2023): This group includes breast cancer patients who were treated at our institution from January 1, 2015, to September 30, 2023, and received immunotherapy or neoadjuvant immunotherapy. Clinical samples (e.g., fresh tissue from diagnostic punctures, residual tumor tissue post-surgery, blood samples, and imaging data) from these patients will be retrospectively collected and analyzed. The data will be used to build and validate the predictive model for immunotherapy efficacy.
  Interventions: Other: Retrospective Data Collection and Analysis
- Cohort (2023-Present): This group includes breast cancer patients treated at our institution starting from October 1, 2023, who are potential candidates for immunotherapy or neoadjuvant immunotherapy. Clinical samples (e.g., fresh tissue from diagnostic punctures, residual tumor tissue post-surgery, blood samples, and imaging data) will be prospectively collected. These samples will undergo multi-omics analysis (proteomics, transcriptomics, metabolomics) and advanced imaging techniques (imaging mass cytometry and spatial transcriptomics) to further refine and validate the predictive model for immunotherapy efficacy.
  Interventions: Other: Retrospective Data Collection and Analysis

INTERVENTIONS:
Other: Retrospective Data Collection and Analysis — This is a retrospective study involving the collection and analysis of existing clinical data from breast cancer patients who received immunotherapy or neoadjuvant immunotherapy between January 1, 2015, and September 30, 2023. No new interventions are administered as part of this study. The data includes diagnostic puncture tissue, residual tumor tissue post-surgery, blood samples, and imaging data. These samples are analyzed using multi-omics approaches (proteomics, transcriptomics, metabolomics) and advanced imaging techniques (imaging mass cytometry and spatial transcriptomics) to build a predictive model for immunotherapy efficacy.

SUMMARY:
This study aims to collect clinical samples from breast cancer patients who have undergone or are expected to undergo immunotherapy at our institution. The samples, including fresh tissue from diagnostic punctures, residual tumor tissue post-surgery, blood samples, and imaging data, will be used to build a predictive model for immunotherapy efficacy. The research will employ proteomics, transcriptomics, metabolomics sequencing, imaging mass cytometry (IMC), and spatial transcriptomics to construct a multi-omics, multi-dimensional (temporal and spatial) model to predict the effectiveness of immunotherapy.

DETAILED DESCRIPTION:
This research will utilize a comprehensive approach by analyzing various types of clinical samples from breast cancer patients treated with immunotherapy. The integration of proteomic, transcriptomic, and metabolomic data, along with advanced imaging techniques like IMC and spatial transcriptomics, will allow for a detailed understanding of the tumor microenvironment and its response to immunotherapy. This multi-dimensional analysis aims to enhance the accuracy of predicting immunotherapy outcomes, thereby aiding in personalized treatment strategies for breast cancer patients. The study adheres strictly to ethical guidelines, ensuring patient confidentiality and welfare are maintained throughout the research process.

ELIGIBILITY:
Inclusion Criteria:

- Female, aged ≥ 18 years.

Pathologically confirmed diagnosis of breast cancer.

Patients who received immunotherapy/neoadjuvant immunotherapy at our institution between January 1, 2015, and September 30, 2023 (retrospective cohort), or patients who may receive immunotherapy/neoadjuvant immunotherapy starting from October 1, 2023 (prospective cohort).

Availability of sufficient tumor tissue samples (e.g., fresh biopsy tissue, residual tumor tissue post-surgery).

Availability of blood samples and imaging data.

Signed informed consent (for the prospective cohort).

Exclusion Criteria:

* Male breast cancer patients.

Inability to provide sufficient tumor tissue samples or other clinical data.

Presence of severe comorbidities (e.g., active infections, severe cardiac, hepatic, or renal dysfunction) that may affect the safety assessment of immunotherapy.

Lack of signed informed consent (for the prospective cohort).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population Description:
  The study population consists of female breast cancer patients who received or are expected to receive immunotherapy/neoadjuvant immunotherapy at our institution. The study is divided into two cohorts:
  Retrospective Cohort (2015-2023): Includes patients who received immunotherapy/neoadjuvant immunotherapy between January 1, 2015, and September 30, 2023.
  Prospective Cohort (2023-Present): Includes patients who may receive immunotherapy/neoadjuvant immunotherapy starting from October 1, 2023.
  All participants are female, aged ≥ 18 years, and able to provide sufficient tumor tissue samples, blood samples, and imaging data.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2027-11-17 (Estimated)

PRIMARY OUTCOMES:
Predictive Accuracy of Immunotherapy Efficacy Model | From the date of sample collection (retrospective cohort: 2015-2023; prospective cohort: 2023-present) until the end of follow-up (up to 5 years post-treatment).
  The primary outcome is the predictive accuracy of the multi-omics and multi-dimensional model in determining the efficacy of immunotherapy in breast cancer patients. The model will be evaluated based on its ability to correctly classify patients as responders or non-responders to immunotherapy using clinical outcomes (e.g., progression-free survival, overall survival) as the gold standard.

SECONDARY OUTCOMES:
Correlation Between Multi-Omics Profiles and Immunotherapy Response | From the date of sample collection until the end of follow-up (up to 5 years post-treatment).
  To assess the relationship between proteomic, transcriptomic, and metabolomic profiles of tumor tissue and the clinical response to immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Wu, Principal Investigator — Hangzhou Institute of Medicine (HIM), Chinese Academy
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Due to ethical and privacy concerns, the individual participant data will not be shared outside the research team.